CLINICAL TRIAL: NCT04290390
Title: A Drug-Drug Interaction Study to Evaluate the Effects of Strong CYP3A Induction and Inhibition on the Pharmacokinetics of Segesterone Acetate and Ethinyl Estradiol From the Annovera™ Contraceptive Vaginal System
Brief Title: Annovera™ Drug-Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TherapeuticsMD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ANNOV3454-2 PMR
Record Dates: First submitted 2020-02-10; First posted 2020-02-28 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Women; Contraception
Keywords: rifampin; itraconazole; CYP3A
MeSH Terms: interventions — segesterone acetate and ethinyl estradiol vaginal system; Rifampin; Itraconazole

STUDY DESIGN:
Intervention Model Description: Two cohort, open label, randomized, two period (Cycle 1 and Cycle 2) crossover study. Subjects may only participate in one randomized sequence of one cohort. Subjects will be assigned to either Cohort 1 (itraconazole) or Cohort 2 (rifampin). Once assigned, a subject will then be randomized to a Sequence Group within the cohort. There will be at least a 4-week washout between Treatment Cycle 1 and Cycle 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Annovera (alone) (Active Comparator): Annovera taken alone (without itraconazole or rifampin)
  Interventions: Drug: Segesterone Acetate and Ethinyl Estradiol
- Annovera with itraconazole use (Active Comparator): Subjects will dose with 200 mg/day of itraconazole for five days before Annovera insertion and through Days 1 to 8 of Annovera use
  Interventions: Drug: Segesterone Acetate and Ethinyl Estradiol; Drug: Itraconazole
- Annovera with rifampin use (Active Comparator): Subjects will dose with 600 mg/day rifampin for 8 days, between Days 4 to 11 of Annovera use during their respective treatment cycles
  Interventions: Drug: Segesterone Acetate and Ethinyl Estradiol; Drug: Rifampin

INTERVENTIONS:
Drug: Segesterone Acetate and Ethinyl Estradiol — Contraceptive Vaginal System
  Other Names: Annovera
Drug: Rifampin — CYP3A inducer
  Arms: Annovera with rifampin use
Drug: Itraconazole — CYP3A inhibitor
  Arms: Annovera with itraconazole use

SUMMARY:
A Drug-Drug Interaction (DDI) study to evaluate the effects of itraconazole and rifampin on the Pharmacokinetics of Segesterone Acetate and Ethinyl Estradiol from the Annovera Contraceptive Vaginal System (CVS)

ELIGIBILITY:
Inclusion Criteria

All of the following criteria must be met for the participants to be eligible for the study:

* a. Healthy women, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening) sterile or at risk of becoming pregnant, inclusive of ages 18 to 35* years at the enrollment visit.
* b. Body Mass Index (BMI) > 18.5 and ≤ 29.0 kg/m2 and body weight ≥ 45.0 kg.
* c. Intact uterus and both ovaries.
* d. Prior history of regular menstrual cycles that usually occur every 28 ± 7 days when not using hormonal contraception; if postpartum or post-abortal, history of regular menstrual cycles of 21 to 35 days in length and resumption of at least one cycle with a cycle length consistent with her past cycles.
* e. In the opinion of the Investigator, able to comply with the protocol, eg, live within the study site catchment area or within a reasonable distance from the study site.
* f. If not sterile and sexually active with a non-sterile male partner, willing to use one of the following acceptable contraceptive methods throughout the study:
* intra-uterine contraceptive device without hormone release system placed at least 28 days prior to the start of the first treatment cycle;
* male condom with intravaginally applied spermicide starting at least 21 days prior to the start of the first treatment cycle;
* g. If not sterile and sexually active with a sterile male partner, the partner is at least 6 months post-vasectomy.
* h. Willing to abstain from Tylenol/acetaminophen use and from consuming grapefruit or grapefruit juice from 7 days pre-dose until after the last PK blood sample collection of each period.
* i. Willing to abstain from alcohol from 24 hours pre-dose until after the last PK blood sample collection of each period.
* j. Signed informed consent prior to entry into the trial.

(*Upper age limit based on normal ovarian changes (ovarian reserve) prevalent in women with advancing age (> 35 years of age) that may alter patterns of follicle development and/or confound interpretations of data regarding patterns of follicle development)

Exclusion Criteria

Contraindications for enrollment will be the same as those for use of CHCs and additional criteria important to the objectives of this study and include:

* a. Known hypersensitivity to estrogens or progestins.
* b. Pregnant, trying to become pregnant, or breastfeeding.
* c. Known hypersensitivity to silicone rubber.
* d. Undiagnosed abnormal vaginal bleeding.
* e. Undiagnosed vaginal discharge, vaginal lesions or abnormalities. Participants diagnosed at screening with a chlamydia or gonococcus infection may be included in the trial following treatment; partner treatment is also recommended. Investigators should make a determination if participants are at high risk for reinfection, eg, multiple sex partners, untreated partner, and whether such participants can be included.
* f. History of pelvic inflammatory disease since the participant's last pregnancy.
* g. History of toxic shock syndrome.
* h. In accordance with the Bethesda system of classification: Women with a current (within the last 20 months) abnormal Papanicolaou smear (Pap smear) suggestive of high-grade pre-cancerous lesion(s), including high grade squamous intraepithelial lesion.
* i. Cystoceles or rectoceles or other anatomical abnormality that would preclude use of a vaginal ring.
* j. Women planning to undergo major surgery during the trial.
* k. Current or past thrombophlebitis or thromboembolic disorders.
* l. History of venous thrombosis or embolism in a first-degree relative, < 55 years of age suggesting a familial defect in the blood coagulation system, which in the opinion of the Principal Investigator (PI), suggests that use of a hormonal contraceptive could pose a significant risk.
* m. Cerebrovascular or cardiovascular disease.
* n. History of retinal vascular lesions, unexplained partial or complete loss of vision.
* o. Known or suspected carcinoma of the breast.
* p. Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia.
* q. Past history of any other carcinoma unless in remission for more than five years.
* r. Current or history of medically diagnosed severe depression, which, in the opinion of the Investigator, could be exacerbated by the use of a hormonal contraceptive.
* s. Has a Type D personality type as assessed by the DS14 test (Standard Assessment of Negative Affectivity, Social Inhibition and Type D Personality).
* t. Headaches with focal neurological symptoms.
* u. Severe constipation in the opinion of the Investigator.
* v. History of cholestatic jaundice of pregnancy or jaundice with prior steroid use.
* w. Benign or malignant liver tumors; active liver disease.
* x. Diastolic blood pressure (BP) > 85 mm Hg and/or systolic BP > 135 mm Hg after 5 to 10 minutes rest (at Screening).
* y. Known or suspected alcoholism or drug abuse within their lifetime, or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine, crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
* z. Elevated serum fasting clinical chemistry values or complete blood count (CBC) values designated clinically significant by the Investigator and/or medically qualified Sub-Investigator.
* aa. Screening hemoglobin levels less than 115 g/L or hematocrit less than 0.32 L/L.
* bb. Participation in another clinical trial involving the administration of an investigational drug or marketed drug or device within the last 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
* cc. Use of liver enzyme inducers on a regular basis and sex steroid hormone treatments (see Section 8.3 for list of exclusionary medications).
* dd. Use of monthly injectable contraceptives, unless suspended 2 months before initiation of the treatment. Use of Depo-Provera® [depot medroxyprogesterone acetate] unless suspended 9 months before treatment.
* ee. Current use of implanted hormonal contraceptives, including Mirena® [progestin containing intrauterine system], Jadelle®, Norplant®, Implanon® or Nexplanon (if now available in the USA).**
* ff. Known HIV, Hepatitis B or Hepatitis C infection.
* gg. History of frequent vaginal infections in the opinion of the Investigator.
* hh. Known hypersensitivity or prior adverse reaction to itraconazole, or to any of the other azoles or to rifampin, or to any of the rifamycins.

(*Women using non-hormonal intrauterine devices are permitted to enroll in the study.) (**Participants using any of the implanted hormonal methods who request removal for reasons unrelated to the purpose of enrollment in this study may be considered for participation.)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Area-under-the-curve (AUC) of rifampin and itraconzaole on Annovera (segesterone acetate and ethinyl estradiol) | Day 1 for itraconazole cohort, Day 11 for rifampin cohort
  AUC for 24 hours for segesterone acetate and ethinyl estradiol
Maximum concentration (Cmax) of rifampin and itraconzaole on Annovera (segesterone acetate and ethinyl estradiol) | Day 1 for itraconazole cohort, Day 11 for rifampin cohort
  Cmax for segesterone acetate and ethinyl estradiol

SECONDARY OUTCOMES:
Safety - Number of Participants with Adverse Events | Screening through 14 days following Annovera removal
  Serious adverse events (SAEs) and adverse events (AEs)
Safety - Vital signs - systolic and diastolic blood pressure | Through study completion, an average of 4 months
  Measurements of systolic and diastolic blood pressure will be compared from Screening to end of treatment/end of study
Safety - Vital signs - pulse | Through study completion, an average of 4 months
  Measurements of pulse will be compared from Screening to end of treatment/end of study
Tolerability -Discontinuation rates | Through study completion, an average of 4 months
  Participant rates of discontinuation due to AEs will provide information regarding tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Mirkin, MD, Study Chair — TherapeuticsMD
Locations (1):
- Syneos Health, Québec, Quebec, Canada